CLINICAL TRIAL: NCT02161874
Title: A Prospective, Randomized-controlled Evaluation of Biomet 3i's T3 Implant System for Integration Success and the Preservation of Crestal Bone
Brief Title: Evaluation of Integration Success and Crestal Bone Preservation Biomet 3i's T3 Implant System
Acronym: OAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3023
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: edentulism; dental implants; clinical study; endosseous; randomized; crestal bone level; T3; Nanotite Certain; Nanotite Certain Prevail; Tapered
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T3 with DCD tapered implant (Experimental): T3 with DCD tapered prevail implant
  Interventions: Device: T3 with DCD tapered Prevail implant
- Nanotite certain tapered implant (Active Comparator): Nanotite Certain tapered implant
  Interventions: Device: Nanotite Certain tapered implant

INTERVENTIONS:
Device: T3 with DCD tapered Prevail implant — T3 with DCD implant with Certain (internal) connection and platform-switch design
  Other Names: T3 with Nanotite; T3 with platform switch
  Arms: T3 with DCD tapered implant
Device: Nanotite Certain tapered implant — Nanotite (DCD) implant with Certain (internal) connection and non- platform-switch design
  Other Names: Nanotite tapered certain; Non-platform switched
  Arms: Nanotite certain tapered implant

SUMMARY:
This study evaluates the T3 implant system for the preservation of alveolar crestal bone and the establishment of initial integration. The new surface-treated features of the implant may contribute to improved soft and hard tissue healing. The success rate of the T3 implant will be no different than that of the control implant, which possess similar geometry but different surface treatments.

DETAILED DESCRIPTION:
This prospective, randomized-controlled study will enroll qualified patients with partial edentulism who will be treated with at least two dental implants. Implant sites will be randomly assigned to receive either a test (T3 implant) or control (Nanotite Certain Tapered implant) with an 80:20 (test:control) randomization ratio.

All implants will be allowed to integrate without occlusal forces and final restorations will be cemented thereafter.

Cumulative success rate and crestal bone regression of both treatment groups will be the primary and secondary study endpoints, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex and any race greater than 18 years of age
* Patients for whom a decision has already been made to use dental implants for the restoration of existing edentulism in the mandible or maxilla.
* Patients must be physically able to tolerate conventional surgical and restorative procedures.
* Patients must agree to be evaluated for each study visit, especially the yearly follow-up visits

Exclusion Criteria:

* Patients with active infection or severe inflammation in the areas intended for implant placement.
* Patients with a > 10 cigarette per day smoking habit.
* Patients with uncontrolled diabetes mellitus.
* Patients with uncontrolled metabolic bone disease where there is a diagnosis of the following: Osteomalacia, primary or secondary hyperparathyroidism, renal osteodystrophy, or Paget's disease of bone.
* Patients with a history of therapeutic radiation to the head
* Patients in need of bone grafting at the site of the intended study implant for augmentation purposes.
* Patients who are known to be pregnant at the screening visit.
* Patients with evidence of severe para-functional habits such as bruxing or clenching.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Cumulative success rate | 1 year
  Implant mobility is assessed by clinical evaluations and correlation to initial placement stability- insertion torque profiles.

SECONDARY OUTCOMES:
Crestal bone changes | 2 years
  Crestal bone regression (amount of bone loss) between the two treatment groups will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Lewis, DMD, Principal Investigator — Eastman Dental Hospital
Locations (4):
- Dr. Tommie VanDeVelde, Antwerp, Belgium
- Dr. Dominique Caspar, Les Bains, France
- Dr. Felix Hanssler, Göppingen, Germany
- Dr. Nicholas Lewis, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No